CLINICAL TRIAL: NCT05012163
Title: Lottery Incentive Nudges to Increase Influenza Vaccinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Geisinger Clinic (Other); Massachusetts Institute of Technology (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0484; P30AG034532 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Influenza; Vaccination; Health Promotion; Health Behavior
Keywords: Lottery; Financial Incentives
MeSH Terms: conditions — Influenza, Human; Health Behavior

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to one of four arms:
  * Pennsylvania Lottery Scratch-Off Financial Incentive
  * Certain Cash Payout Financial Incentive
  * Reminder / Active Control Arm (No Financial Incentive)
  * No Treatment Control Arm
Who Masked: Care Provider
Masking Description: Providers who prescribe vaccination and diagnose conditions will not be randomized to study arms or informed of patient assignment. Although patients will not be explicitly informed of which arm they were randomized to, they will be aware of the messages they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pennsylvania (PA) Lottery Scratch-Off Financial Incentive (Experimental): Participants in this arm will receive a message stating that they will receive a PA lottery $1 scratch-off ticket if they get a flu shot at an upcoming appointment. The message will mention that they could win $5,000 (the top prize for the scratch-off game).
  Note: $1 scratch-off products vary over time; at study implementation, an active game with top prize of $5,000 (or the next-highest top prize) will be selected and will define the prize in the raffle absent upfront odds
  Interventions: Behavioral: Reminder; Behavioral: Financial incentive; Behavioral: Lottery
- Certain Cash Payout Financial Incentive (Experimental): Participants in this arm will receive a message stating that they will receive $1 in cash if they get a flu shot at an upcoming appointment.
  Interventions: Behavioral: Reminder; Behavioral: Financial incentive
- Reminder / Active Control (No Financial Incentive) (Experimental): Participants in this arm will receive a message stating that they can get a flu shot at an upcoming appointment. These participants will not be offered a financial incentive for getting a flu shot.
  Interventions: Behavioral: Reminder
- No Treatment Control (No Intervention): No additional contact beyond standard Geisinger flu shot communications

INTERVENTIONS:
Behavioral: Reminder — Letter, short message service (SMS) text, phone, and/or email
  Arms: Certain Cash Payout Financial Incentive; Pennsylvania (PA) Lottery Scratch-Off Financial Incentive; Reminder / Active Control (No Financial Incentive)
Behavioral: Financial incentive — Letter, SMS, phone, and/or email
  Arms: Certain Cash Payout Financial Incentive; Pennsylvania (PA) Lottery Scratch-Off Financial Incentive
Behavioral: Lottery — Letter, SMS, phone, and/or email
  Arms: Pennsylvania (PA) Lottery Scratch-Off Financial Incentive

SUMMARY:
In the current study, the study team will explore whether small incentives are effective at promoting flu vaccine uptake. The study is designed to compare the relative efficacy of incentives of equal perceived expected value (EV) or equal implementation costs, to assess whether people are more likely to get vaccinated in response to lotteries with very high payoffs than to small certain cash payout or slightly higher-probability, more moderate payoffs. In particular, given the potential appeal of official state lottery tickets, one study arm will receive a Pennsylvania scratch-off lottery ticket for getting a flu vaccine. A primary hypothesis is that lotteries will outperform simple reminders (encouraging respondents to get the flu shot at their upcoming appointment) and the standard of care, representing the ambient healthcare system and public health campaigns to increase vaccination.

DETAILED DESCRIPTION:
During the 2021-22 flu season, the study team will contact Geisinger patients who have a primary care or specialist appointment scheduled during flu season and encourage them to get a flu shot.

Patients will be randomized into 4 to 9 study arms, depending on a sample size projection completed in August 2021. Arms will test the relative efficacy of a variety of small monetary incentives on flu shot uptake. Incentives may include (a) a $1 Pennsylvania scratch-off lottery ticket (with top prize of $5,000), (b) $1 in cash, (c) entry into a raffle for $5,000 absent upfront odds, (d) entry into a raffle for $5,000, with 1-in-5,000 odds of winning, (d) entry into a raffle for $50, with 1-in-50 odds of winning, and (e) entry into a raffle for $500, with 1-in-500 odds of winning. There will be one no-contact control arm and at least 1 reminder control arm (with additional control arms added given sufficient sample size and additional message versions to be tested).

Included in the study will be current Geisinger patients 18+ years of age with no contraindications for flu vaccine who have an appointment scheduled during the study period with a provider who can administer the vaccine. The primary study outcomes will be the rates of flu vaccination and flu diagnosis during the 2021-22 season by targeted patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Pennsylvania mailing address listed
* Geisinger primary care provider (PCP) assigned
* Upcoming appointment with PCP or select specialist who stocks and can administer the vaccine during the study period

Exclusion Criteria:

* Has opted out of receiving messages from Geisinger on all modalities being tested

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57581 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle N Meyer, PhD JD, Principal Investigator — Geisinger Clinic; Christopher F Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date or within 12 months of the primary completion date (whichever comes first). Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: https://osf.io/ahmf2/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pennsylvania (PA) Lottery Scratch-Off Financial Incentive: Participants in this arm will receive a message stating that they will receive a PA lottery $1 scratch-off ticket if they get a flu shot at an upcoming appointment. The message will mention that they could win $5,000 (the top prize for the scratch-off game).
  Note: $1 scratch-off products vary over time; at study implementation, an active game with top prize of $5,000 (or the next-highest top prize) will be selected and will define the prize in the raffle absent upfront odds
  Reminder: Letter, short message service (SMS) text, phone, and/or email
  Financial incentive: Letter, SMS, phone, and/or email
  Lottery: Letter, SMS, phone, and/or email
Period: Overall Study
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Started | 14394 | 14394 | 14394 | 14399
Completed | 14394 | 14394 | 14393 | 14398
Not Completed | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control | Total
Number analyzed (Participants) | 14394 | 14394 | 14394 | 14399 | 57581
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 1 | 1 | 2
  18-65 | 11051 | 11105 | 11097 | 11066 | 44319
  65+ | 3343 | 3289 | 3296 | 3332 | 13260
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8370 | 8306 | 8313 | 8344 | 33333
  Male | 6024 | 6088 | 6081 | 6055 | 24248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 643 | 659 | 701 | 661 | 2664
  Not Hispanic or Latino | 13670 | 13649 | 13624 | 13656 | 54599
  Unknown or Not Reported | 81 | 86 | 69 | 82 | 318
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 42 | 29 | 30 | 29 | 130
  Asian | 135 | 112 | 130 | 148 | 525
  Black or African American | 595 | 609 | 615 | 595 | 2414
  Native Hawaiian or Other Pacific Islander | 50 | 51 | 56 | 53 | 210
  White | 13459 | 13484 | 13448 | 13457 | 53848
  Unknown | 113 | 109 | 115 | 117 | 454

OUTCOME MEASURES:

1. Primary Outcome: Flu Vaccination at Appointment
Description: Received flu vaccination at relevant PCP or specialty appointment.
Time Frame: 3 days after patient is randomized
Population: All enrolled patients were included in analyses, except the two patients who were inadvertently enrolled at age 17.
Measure: Count of Participants; unit: Participants
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Number analyzed (Participants) | 14394 | 14394 | 14393 | 14398
Participants
  No Shot at Appointment | 10461 | 10511 | 10394 | 10746
  Shot at Appointment | 3933 | 3883 | 3999 | 3652
Statistical Analysis 1: Comparison: Pennsylvania (PA) Lottery Scratch-Off Financial Incentive vs Certain Cash Payout Financial Incentive; Null hypothesis: There is no difference in vaccination rates between patients sent messages offering a scratch-off lottery ticket and patients sent messages offering $1 cash in exchange for vaccination; Alternative hypothesis: the vaccination rate is higher in patients sent messages offering scratch-off tickets compared to those sent messages offering $1 cash; Test type: Superiority; p = .506, Regression, Linear — Pairwise comparisons between patients offered scratch-off tickets for vaccination and those in other arms (Analyses 1, 2 and 3) were analyzed in the same regression
Statistical Analysis 2: Comparison: Pennsylvania (PA) Lottery Scratch-Off Financial Incentive vs Reminder / Active Control (No Financial Incentive); Null hypothesis: There is no difference in vaccination rates between patients sent messages offering a scratch-off lottery ticket in exchange for vaccination and those sent active control messages; Alternative hypothesis: the vaccination rate is higher in patients sent messages offering scratch-off tickets compared to those sent active control messages; Test type: Superiority; p = 0.378, Regression, Linear — Comments: Pairwise comparisons between patients offered scratch-off tickets for vaccination and those in other arms (Analyses 1, 2 and 3) were analyzed in the same regression
Statistical Analysis 3: Comparison: Pennsylvania (PA) Lottery Scratch-Off Financial Incentive vs No Treatment Control; Null hypothesis: There is no difference in vaccination rates between patients sent messages offering a scratch-off lottery ticket in exchange for vaccination and those sent no study messages; Alternative hypothesis: the vaccination rate is higher in patients sent messages offering scratch-off tickets compared to those who were not sent messages; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Reminder / Active Control (No Financial Incentive) vs No Treatment Control; Null hypothesis: There is no difference in vaccination rates between patients sent active control messages and those sent no study messages; Alternative hypothesis: the vaccination rate is higher in patients sent active control messages compared to those who were not sent messages; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 5: Comparison: Certain Cash Payout Financial Incentive vs Reminder / Active Control (No Financial Incentive); Null hypothesis: There is no difference in vaccination rates between patients sent messages offering $1 cash in exchange for vaccination and those sent active control messages; Alternative hypothesis: the vaccination rate is higher in patients sent messages offering $1 cash compared to those sent active control messages; Test type: Superiority — Pairwise comparisons between patients offered cash for vaccination and those in active or passive control (Analyses 5 and 6) were analyzed in the same regression; p = .121, Regression, Linear
Statistical Analysis 6: Comparison: Certain Cash Payout Financial Incentive vs No Treatment Control; Null hypothesis: There is no difference in vaccination rates between patients sent messages offering $1 cash in exchange for vaccination and those sent no study messages; Alternative hypothesis: the vaccination rate is higher in patients sent messages offering $1 cash compared to those who were not sent messages; Test type: Superiority; p = .002, Regression, Linear — Pairwise comparisons between patients offered cash for vaccination and those in active or passive control (Analyses 5 and 6) were analyzed in the same regression

2. Secondary Outcome: Flu Vaccination Within 7 Days
Description: Received flu vaccination
Time Frame: Within 7 days of when patient is randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Number analyzed (Participants) | 14394 | 14394 | 14393 | 14398
Participants
  No Shot Within 7 Days | 10119 | 10104 | 10007 | 10343
  Shot Within 7 Days | 4275 | 4290 | 4386 | 4055

3. Secondary Outcome: Flu Diagnosis
Description: Received a "high confidence flu" diagnosis (with positive polymerase chain reaction [PCR]/antigen/molecular test) and/or "likely flu" diagnosis (as assessed via International Classification of Disease [ICD] codes or Tamiflu administration or positive PCR/antigen/molecular test)
  Note that "likely flu" is a superset of the "high confidence flu" diagnoses.
Time Frame: During the 2021-22 flu season (Up to 8 months, from the time the patient is randomized through April 30, 2022)
Measure: Count of Participants; unit: Participants
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Number analyzed (Participants) | 14394 | 14394 | 14393 | 14398
Participants
  No flu diagnosis | 14277 | 14262 | 14298 | 14265
  Flu diagnosis | 117 | 132 | 95 | 133

4. Secondary Outcome: Flu Complications
Description: Diagnosed with flu-related complications
Time Frame: During the 2021-22 flu season (Up to 11 months, from the time the patient is randomized through July 31, 2022)
Measure: Count of Participants; unit: Participants
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Number analyzed (Participants) | 14394 | 14394 | 14393 | 14398
Participants
  No flu complications | 12537 | 12613 | 12593 | 12605
  Flu complications | 1857 | 1781 | 1800 | 1793

5. Other Pre Specified Outcome: Flu Vaccination (Among Subject Cohabitants) Within 28 Days
Description: Cohabitant of study subject received flu vaccination
Time Frame: Within 28 days of when the study subject is randomized
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Flu Vaccination at Appointment by Gender
Description: Received flu vaccination at relevant PCP or specialty appointment.
Time Frame: 3 days after the patient is randomized.
Population: All enrolled patients were included in analyses, except the two patients who were inadvertently enrolled at age 17.
Measure: Count of Participants; unit: Participants
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Number analyzed (Participants) | 14394 | 14394 | 14393 | 14398
Participants
  Female: number analyzed (Participants) | 8370 | 8306 | 8312 | 8344
  Female: No Shot at Appointment | 6207 | 6132 | 6106 | 6290
  Female: Shot at Appointment | 2163 | 2174 | 2206 | 2054
  Male: number analyzed (Participants) | 6024 | 6088 | 6081 | 6054
  Male: No Shot at Appointment | 4254 | 4379 | 4288 | 4456
  Male: Shot at Appointment | 1770 | 1709 | 1793 | 1598

7. Other Pre Specified Outcome: Flu Vaccination at Appointment by Race
Description: Received flu vaccination at relevant PCP or specialty appointment.
Time Frame: 3 days after the patient is randomized.
Population: All enrolled patients were included in analyses, except the two patients who were inadvertently enrolled at age 17.
Measure: Count of Participants; unit: Participants
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Number analyzed (Participants) | 14394 | 14394 | 14393 | 14398
Participants
  American Indian or Alaska Native: number analyzed (Participants) | 42 | 29 | 30 | 29
  American Indian or Alaska Native: No Shot at Appointment | 33 | 23 | 18 | 21
  American Indian or Alaska Native: Shot at Appointment | 9 | 6 | 12 | 8
  Asian: number analyzed (Participants) | 135 | 112 | 130 | 148
  Asian: No Shot at Appointment | 92 | 78 | 89 | 101
  Asian: Shot at Appointment | 43 | 34 | 41 | 47
  Black or African American: number analyzed (Participants) | 595 | 609 | 615 | 595
  Black or African American: No Shot at Appointment | 496 | 521 | 509 | 515
  Black or African American: Shot at Appointment | 99 | 88 | 106 | 80
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 50 | 51 | 56 | 53
  Native Hawaiian or Other Pacific Islander: No Shot at Appointment | 37 | 42 | 36 | 37
  Native Hawaiian or Other Pacific Islander: Shot at Appointment | 13 | 9 | 20 | 16
  Unknown: number analyzed (Participants) | 113 | 109 | 115 | 117
  Unknown: No Shot at Appointment | 85 | 90 | 93 | 96
  Unknown: Shot at Appointment | 28 | 19 | 22 | 21
  White: number analyzed (Participants) | 13459 | 13484 | 13447 | 13456
  White: No Shot at Appointment | 9718 | 9757 | 9649 | 9976
  White: Shot at Appointment | 3741 | 3727 | 3798 | 3480

8. Other Pre Specified Outcome: Flu Vaccination at Appointment by Ethnicity
Description: Received flu vaccination at relevant PCP or specialty appointment.
Time Frame: 3 days after the patient is randomized.
Population: All enrolled patients were included in analyses, except the two patients who were inadvertently enrolled at age 17.
Measure: Count of Participants; unit: Participants
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
Number analyzed (Participants) | 14394 | 14394 | 14393 | 14398
Participants
  Hispanic or Latino: number analyzed (Participants) | 643 | 659 | 700 | 660
  Hispanic or Latino: No Shot at Appointment | 511 | 517 | 525 | 530
  Hispanic or Latino: Shot at Appointment | 132 | 142 | 175 | 130
  Not Hispanic or Latino: number analyzed (Participants) | 13670 | 13649 | 13624 | 13656
  Not Hispanic or Latino: No Shot at Appointment | 9889 | 9922 | 9812 | 10153
  Not Hispanic or Latino: Shot at Appointment | 3781 | 3727 | 3812 | 3503
  Unknown: number analyzed (Participants) | 81 | 86 | 69 | 82
  Unknown: No Shot at Appointment | 61 | 72 | 57 | 63
  Unknown: Shot at Appointment | 20 | 14 | 12 | 19

ADVERSE EVENTS:
Description: This is a minimal risk study, and has received expedited IRB review in keeping with 45 CFR §46.110. EHR and claims data will report inputs (i.e., the subject's assigned arm) and outcomes (i.e., flu vaccination, flu diagnosis, flu-like symptoms). We therefore did not monitor the data for AE/SAEs.
Arm/Group | Pennsylvania (PA) Lottery Scratch-Off Financial Incentive | Certain Cash Payout Financial Incentive | Reminder / Active Control (No Financial Incentive) | No Treatment Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT05012163/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT05012163/SAP_001.pdf